CLINICAL TRIAL: NCT00408850
Title: Mechanisms of Sympathetic Overactivity in the Metabolic Syndrome: Effects of Reversing Insulin Resistance by Drug Treatment
Brief Title: Effects of Pioglitazone Treatment on Sympathetic Nervous System Function in Metabolic Syndrome Obesity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baker Heart Research Institute (Other)
Collaborators: National Heart Foundation, Australia (Other)
Responsible Party: Principal Investigator, Nora E. Straznicky, Dr, Baker Heart Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G 06M 2610
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Metabolic Syndrome
Keywords: sympathetic nervous system, pioglitazone, metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Pioglitazone; Sugars; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Active Comparator): pioglitazone 15 mg for 6 weeks followed by 30 mg for 6 weeks
  Interventions: Drug: Pioglitazone
- sugar pill (Placebo Comparator): Placebo comparator
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Pioglitazone — 15 mg per day for 6 weeks and 30 mg per day for further 6 weeks
  Other Names: Actos
  Arms: Pioglitazone
Drug: sugar pill — One capsule daily for 6 weeks followed by two capsules per day for next 6 weeks
  Other Names: Lactose
  Arms: sugar pill

SUMMARY:
An abdominal distribution of fat is associated with the greatest heart disease risk, because commonly, several risk factors of metabolic origin cluster in these individuals. When this occurs the condition is called the 'metabolic syndrome'.

Increased activity of the sympathetic nervous system resulting in enhanced release of the stress hormone 'noradrenaline', may be one mechanism by which adverse cardiovascular and metabolic sequela of the metabolic syndrome might be mediated. Impaired insulin action may be one factor contributing to increased noradrenaline release.

The aim of this Study is to determine whether treatment with a drug called pioglitazone which is known to improve insulin action, results in reduced sympathetic nervous system activity and stress hormone release when compared to treatment with a dummy drug (placebo).

DETAILED DESCRIPTION:
The rapidly growing burden of obesity together with a population that is becoming older raises the importance of effective strategies for the primary prevention and treatment of the metabolic syndrome in order to combat the epidemic of type 2 diabetes and to reduce the increased risk of cardiovascular mortality.

Increased sympathetic nervous system activity may participate in the pathogenesis and complications of the metabolic syndrome. This Study will use a randomised controlled design to evaluate the effects of pioglitazone treatment on sympathetic activity in middle-aged subjects with the metabolic syndrome.The results will generate new information on the neuroadrenergic effects of thiazolidinediones in this clinical setting. This is relevant to the understanding of the pathophysiology of the metabolic syndrome and to its clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 45-65 years,
* non-smokers,
* HOMA index > 2.5 and
* who meet ATP III criteria for the metabolic syndrome

Exclusion Criteria:

* History of diabetes,
* previous MI, stroke, heart failure, impaired hepatic or renal function.
* Inability to cease medications which may affect study parameters.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Sympathetic nervous system activity, measured as muscle sympathetic nervous activity and whole-body noradrenaline spillover | 12 weeks treatment

SECONDARY OUTCOMES:
Baroreflex function, adrenoceptor expression | 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nora E Straznicky, PhD, MPH, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Baker Heart Research Institute, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Esler M, Straznicky N, Eikelis N, Masuo K, Lambert G, Lambert E. Mechanisms of sympathetic activation in obesity-related hypertension. Hypertension. 2006 Nov;48(5):787-96. doi: 10.1161/01.HYP.0000242642.42177.49. Epub 2006 Sep 25. No abstract available. PMID 17000932
- [Background] Straznicky NE, Lambert EA, Lambert GW, Masuo K, Esler MD, Nestel PJ. Effects of dietary weight loss on sympathetic activity and cardiac risk factors associated with the metabolic syndrome. J Clin Endocrinol Metab. 2005 Nov;90(11):5998-6005. doi: 10.1210/jc.2005-0961. Epub 2005 Aug 9. PMID 16091482
- [Derived] Straznicky NE, Grima MT, Sari CI, Lambert EA, Phillips SE, Eikelis N, Kobayashi D, Hering D, Mariani JA, Dixon JB, Nestel PJ, Karapanagiotidis S, Schlaich MP, Lambert GW. Reduction in peripheral vascular resistance predicts improvement in insulin clearance following weight loss. Cardiovasc Diabetol. 2015 Aug 22;14:113. doi: 10.1186/s12933-015-0276-2. PMID 26297500
- [Derived] Straznicky NE, Grima MT, Sari CI, Eikelis N, Lambert GW, Nestel PJ, Richards K, Dixon JB, Schlaich MP, Lambert EA. Pioglitazone treatment enhances the sympathetic nervous system response to oral carbohydrate load in obese individuals with metabolic syndrome. Metabolism. 2015 Jul;64(7):797-803. doi: 10.1016/j.metabol.2015.03.006. Epub 2015 Mar 18. PMID 25827058
- [Derived] Straznicky NE, Grima MT, Lambert EA, Sari CI, Eikelis N, Nestel PJ, Phillips SE, Hering D, Karapanagiotidis S, Dixon JB, Schlaich MP, Lambert GW. Arterial norepinephrine concentration is inversely and independently associated with insulin clearance in obese individuals with metabolic syndrome. J Clin Endocrinol Metab. 2015 Apr;100(4):1544-50. doi: 10.1210/jc.2014-3796. Epub 2015 Jan 15. PMID 25590214
- [Derived] Straznicky NE, Grima MT, Sari CI, Eikelis N, Lambert GW, Nestel PJ, Karapanagiotidis S, Wong C, Richards K, Marusic P, Dixon JB, Schlaich MP, Lambert EA. A randomized controlled trial of the effects of pioglitazone treatment on sympathetic nervous system activity and cardiovascular function in obese subjects with metabolic syndrome. J Clin Endocrinol Metab. 2014 Sep;99(9):E1701-7. doi: 10.1210/jc.2014-1976. Epub 2014 Jun 17. PMID 24937541